CLINICAL TRIAL: NCT05812092
Title: A Prospective Clinical/Radiological Outcome Study of the CONDUIT™ Interbody Cervical System With Supplemental Fixation for the Treatment of One and/or Two Level Cervical Degenerative Disc Disease and/or Cervical Spinal Instability
Brief Title: Treatment of One and/or Two Level Cervical Degenerative Disc Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Research Source (Network)
Responsible Party: Sponsor
Other Study IDs: ONRI-OP-001
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- DePuy Synthes Cervical Plating System: All enrolled patients will receive CONDUIT Interbody Cervical System with supplemental fixation using a DePuy Synthes Cervical Plating System.
  Interventions: Device: CONDUIT Interbody Cervical System with DePuy Synthes Cervical Plating System

INTERVENTIONS:
Device: CONDUIT Interbody Cervical System with DePuy Synthes Cervical Plating System — CONDUIT Interbody Cervical System will be inserted between C2 through T1 and fixated using a DePuy Synthes Cervical Plating System at 1 or 2 levels.

SUMMARY:
The objective of this study is to collect clinical and radiographic outcomes using the CONDUIT™ Interbody Cervical System with supplemental fixation using a DePuy Synthes Cervical Plating System.

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate the performance of the CONDUITTM Interbody Cervical System in reducing pain and degree of disability as measured using the Neck Disability Index (NDI). Recruitment will occur from the patient population of the investigator. All patients will be evaluated for participation in the study by using the inclusion/exclusion listed below. Subjects need to meet all the inclusion and none of the exclusion. The responsibility is exclusively maintained by the investigator of any potential study participant as defined by the inclusion/ exclusion. Patients will consent to participating in the study, prior to any study procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject; at least 18 years of age
2. Diagnosis of radiculopathy or myelopathy with radiculopathy of the cervical spine, with pain, paresthesias or paralysis in a specific nerve root distribution C2 through T1, including at least one of the following:

   1. Neck and/or arm pain of at least 30/100 mm on the visual analogue scale (VAS) scale
   2. Decreased muscle strength of at least one level on the clinical evaluation (0 to 5) scale
   3. Abnormal sensation including hyperesthesia or hypoesthesia; and/or
   4. Abnormal reflexes
3. Symptomatic cervical disc disease, facet arthropathy, or cervical spinal stenosis at 1 or 2 levels between C2 and T1, suitable for treatment with anterior discectomy, decompression, and fusion
4. Radiographically determined pathology at the level to be treated correlating to primary symptoms including at least one of the following:

   1. Decreased disc height on radiography,) in comparison to a normal adjacent disc
   2. Degenerative spondylosis
   3. Disc herniation
5. NDI Score >30%.
6. Unresponsive to non-operative, conservative treatment (rest, heat, electrotherapy, physical therapy, chiropractic care and/or analgesics) for:

   1. Approximately six weeks from radiculopathy or myelopathy with radiculopathy symptom onset; or
   2. Have the presence of symptoms or signs of nerve root/spinal cord compression despite continued non-operative, conservative treatment; or
   3. Sooner than 6 weeks for worsening symptoms of neurologic compromise.
7. Reported to be medically cleared for surgery.
8. Physically and mentally able and willing to comply with the Protocol, including the ability to read and complete required forms and willing and able to adhere to the scheduled follow-up visits and requirements of the Protocol.
9. Signed informed consent provided by subject.

Exclusion Criteria:

1. Have an active systemic infection or infection at the operative site.
2. Have a history of or anticipated treatment for active systemic infection, including HIV or Hepatitis C.
3. Have previous trauma to the C2 to T1 levels resulting in significant bony or disco- ligamentous cervical spine injury.
4. Have had any prior spine surgery at the operative level(s).
5. Have osteoporosis
6. Have Paget's disease of bone, osteomalacia or any other metabolic bone disease other than osteoporosis (addressed above).
7. Have active malignancy that included a history of any invasive malignancy (except non- melanoma skin cancer),unless the subject had been treated with curative intent and there had been no clinical signs or symptoms of the malignancy for at least five years.
8. Have symptomatic cervical disc disease or significant cervical spondylosis at more than 2 levels.
9. Have a known allergy to titanium.
10. Are currently pregnant or breastfeeding at time of enrollment or have plans to become pregnant within the next three years.
11. Have rheumatoid arthritis, lupus, or other autoimmune disease affecting the musculoskeletal system
12. Have diseases or conditions that would preclude accurate clinical evaluation in the opinion of the Investigator
13. Have concomitant conditions requiring daily, high-dose oral and/or inhaled steroids.

    High dose steroid use is defined as:
    1. Daily, chronic use of oral steroids equivalent to 5 mg/day of prednisone or greater.
    2. Daily, chronic use of inhaled corticosteroids (at least twice per day).
    3. Use of short-term (less than 10 days) oral steroids at a daily dose greater than 40mg prednisone equivalent within one month of the study procedure.
14. Have current or recent history (within 1 year prior to screening) of substance abuse (alcoholism and/or narcotic addiction) requiring intervention.
15. Have a Body Mass Index (BMI) > 40 kg/m2.
16. Taking medications known to potentially interfere with bone/soft tissue healing (e.g., high-dose oral and/or inhaled steroids, immunosuppressant medication, chemotherapeutic agents). High dose steroid use as defined in Exclusion Criterion 13.
17. Have pending personal litigation relating to spinal injury (worker's compensation is not an exclusion).
18. Have a current history of heavy smoking (more than one pack of cigarettes per day).
19. Currently reside in a location, or anticipating a potential relocation, that may interfere with completion of follow-up examinations.
20. Have mental illness or belonged to a vulnerable population, as determined by the investigator (e.g., prisoner or developmentally disabled), that would compromise ability to provide informed consent or compliance with follow-up requirements.
21. Have an uncontrolled seizure disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male or female subject; at least 18 years of age. Diagnosis of radiculopathy or myelopathy with radiculopathy of the cervical spine, with pain, paresthesias or paralysis in a specific nerve root distribution C2 through T1.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure: | 12 months
  Number of participants with a 15% improvement in NDI score (based on 100% scale) compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- DFW Center for Spinal Disorders, Fort Worth, Texas, United States